CLINICAL TRIAL: NCT07007897
Title: Toric Alignment Observational Study 2025-1
Brief Title: Observational Study - TA- 2025-1
Acronym: TA OS 2025-1
Status: Enrolling by invitation | Type: Observational
Sponsor: Haag-Streit AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 9360002
Record Dates: First submitted 2025-03-17; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Optical Biometry — Biometric measurements of the eye used for surgical planning will be obtained.
Procedure: Cataract Surgery — A video recording of the surgical procedure will be obtained.

SUMMARY:
This multi-centric, prospective observational study collects biometric datasets as well as associated video recordings of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cataracts (any grade),
* Seeking cataract treatment,
* willing to provide informed consent.

Exclusion Criteria:

* Active ocular infections or trauma.
* Poor fixation ability (e.g., severe nystagmus).
* Prior intraocular surgery.
* Seeking toric IOL implantation requiring ink marking.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual over the age of 21 seeking elective cataract surgery at the study sites.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biometric data | one-time measurement before surgery
  collect anonymised biometric data from patients undergoing elective cataract surgery
Video recording | during the surgical procedure
  collect anonymised video recording of surgical procedure from patients undergoing elective cataract surgery

SECONDARY OUTCOMES:
Software algorith | up to 6 months
  Verification of software algorithms that use the biometric data to analyse the video recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Rübel, PhD, Study Chair — Haag-Streit; Julian V Kool van Langenberghe, ing, Study Director — Haag-Streit
Locations (2):
- United States (2):
  - East Valley Ophthalmology, Mesa, Arizona
  - Pacific Clear Vision Institute, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT07007897/ICF_000.pdf